CLINICAL TRIAL: NCT04622072
Title: A Single-arm, Open, Multi-center Phase I/II Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Effectiveness of XZP-5809-TT1 Tablets in Patients With T790M Mutation-positive Locally Advanced or Metastatic Non-small Cell Lung Cancer Who Have Progressed After Treatment With Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFR-TKI).
Brief Title: XZP-5809-TT1 Tablets in Patients With T790M Mutation-positive Locally Advanced or Metastatic Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: Sihuan Pharmaceutical Holdings Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XZP-5809-TT1-1001
Record Dates: First submitted 2020-10-13; First posted 2020-11-09 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2021-05

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): For dose escalation phase, subjects are enrolled for different doses of the experimental drug.
  Interventions: Drug: XZP-5809-TT1 Tablet

INTERVENTIONS:
Drug: XZP-5809-TT1 Tablet — Single tartrate of XZP-5809

SUMMARY:
The trial is divided into two parts, one is dose escalation phase, the second one is dose expansion phase.

For dose escalation phase, the main purpose is to evaluate safety and tolerability of XZP-5809-TT1 tablets after treatment with epidermal growth factor receptor tyrosine kinase inhibitor (EGFR-TKI) in patients With T790M Mutation-positive Locally Advanced or Metastatic Non-small Cell Lung Cancer, and to determine the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT).

For dose expansion phase, the main purpose is to evaluate Objective response rate (ORR) in patients With T790M Mutation-positive Locally Advanced or Metastatic Non-small Cell Lung Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced or metastatic NSCLC who are diagnosed by histology or cytology and are not suitable for surgery or radiotherapy;
* Patients with EGFR sensitive mutations (including deletion of exon 19, L858R mutation of exon 21, at least one of the above mutations) And after the last treatment (regardless of TKI or chemotherapy), the tissue/cytology specimens collected have been passed through a tertiary A hospital or confirmed as T790M+ by the central laboratory;
* The patient's disease progression after the first or/and second-generation EGFR-TKIs treatment (with imaging or pathological evidence, judged by the research center);
* Life expectancy is not less than 12 weeks, ECOG(Eastern Cooperative Oncology Group, ECOG score) is as follows:

ECOG score in the dose-escalation phase: 0~1 points, and no deterioration within 2 weeks before enrollment, ECOG score during dose expansion stage: 0~2 points, and no deterioration within 2 weeks before enrollment;

* According to RECIST 1.1, the patient has at least one imaging (CT/MRI) measurable lesion. When the patient has at least one baseline Tumor lesions meet the following requirements: accurate measurement at baseline, non-lymph node lesions with longest diameter ≥10 mm, or short diameter ≥15 mm Of lymph node lesions. Have not received local treatments such as radiotherapy in the past, and have not been used for research screening biopsy (if there is only one Measurable lesions, biopsy of the lesions is allowed, but the lesions must be performed at least 14 days after the screening biopsy Baseline imaging examination), the measurement method is computed tomography [CT] or magnetic resonance imaging [MRI]);
* The organ function level must meet the following requirements (no blood transfusion or blood products, no use of hematopoietic stimulating factors, No albumin or blood products are used): absolute neutrophil count (ANC) ≥1.5×109/L, platelet count (PLT)

  ≥75×109/L, hemoglobin (Hb) ≥90 g/L; serum total bilirubin ≤1.5 times the upper limit of normal, aspartate aminotransferase (AST) And alanine aminotransferase (ALT) ≤2.5 times the upper limit of normal value (if there is liver metastasis, total bilirubin ≤3 times the upper limit of normal value is allowed, AST, ALT≤5 times the upper limit of normal); Creatinine clearance (Ccr) ≥50 ml/min (according to Cockcroft and Gault formula); Note: If the researcher thinks it is necessary to retest (the reason for the retest must be recorded), the above laboratory examination can only be retested once. complex After the test meets the standard, then the laboratory parameters can be considered qualified.
* Premenopausal women who are likely to have children must have a pregnancy test within 7 days before starting treatment, and the pregnancy test must be negative Sex, must be non-lactating period; infertile women can not take pregnancy test and contraception, but must meet: age 50 Over the age of, not using hormone therapy and menopause for at least 12 months, or have been sterilized. All enrolled patients (regardless of male (Sexual or female) should take adequate barrier contraceptive measures during the entire treatment period and 3 months after the end of treatment;
* Volunteer to join the group and sign the informed consent, follow the trial treatment plan and visit plan.

Exclusion Criteria:

* Have received any of the following treatments in the past:

  1. First medication (first medication refers to the first use of the test drug, hereinafter referred to as the first medication) patient use within 6 weeks Have used nitrosoureas or mitomycin C, or have used other cytotoxic chemotherapeutics or their drugs within 3 weeks before the first administration His anti-cancer drugs;
  2. The time from receiving any EGRF-TKI treatment to the first dose does not exceed the 5 half-life of the drug (for example, Elotinib is not more than 8 days, gefitinib is not more than 10 days, icotinib is not more than 2 days, and afatinib is not more than 8 days day);
  3. The time from receiving other experimental drugs or analogues to the first dose does not exceed the drug's 5 half-life or 14 days (whichever Senior citizens);
  4. The time from receiving other immune preparations to the first administration does not exceed 28 days;
  5. Major surgery (excluding vascular access establishment surgery and biopsy surgery) within 4 weeks before the first medication;
  6. The patient has received more than 30% bone marrow radiotherapy or large-area irradiation (excluding bone transfer) within 4 weeks before the first medication.
* Have used third-generation EGFR-TKI drugs, including but not limited to osimertinib mesylate (Teresa®), Rociletinib (CO-1686), Olmutinib (Olita®, HM61713), ASP8273, EGF816, Ametidine mesylate Ni, Iflutinib mesylate (AST2818), Maihuatinib, Ivitinib, etc. or the raw materials and generic drugs of these drugs;
* CYP3A4 strong inhibitors or strong inducers have been used within 7 days before the first administration; CYP3A4 strong inhibitors or strong inducers have been used within 14 days before the first administration Anti-tumor medicines and Chinese medicine preparations, Chinese medicines and Chinese medicine preparations with tumor adjuvant treatment effects, and exclusion criteria Standard 1) Other drugs with anti-tumor activity not mentioned;
* At the beginning of the first medication, there are still unhealed toxic reactions in the previous treatment, and "General Terminology Standards for Adverse Events (CTCAE 5.0)" If the grade exceeds grade 1 (except for hair loss), neuropathy related to previous platinum therapy can be relaxed to grade 2.
* Spinal cord compression or brain metastasis, but the following conditions are allowed to be selected: asymptomatic, stable disease, no need to use before the start of research treatment Patients who have been treated with steroids for 4 weeks (if the brain metastases have received radiotherapy or/and surgery, the radiotherapy and surgery must be separated from the first use1 month and above before medication);
* There are any clinical evidences that suggest severe or uncontrolled systemic diseases, for example, the researcher believes that the patient is not suitable for participation or those that will affect patients' compliance with the research protocol, such as patients with uncontrolled hypertension, patients with uncontrolled diabetes, patients with coronary artery stenosis, patients with aortic dissection, patients with aortic aneurysms, patients with active bleeding Individuals who are on anti-infection treatment;
* Currently existing hepatitis B (hepatitis B surface antigen [HbsAg] positive or core antibody [HbcAb] positive and HBV (hepatitis B virus DNA) positive), hepatitis C (HCV antibody positive and HCV RNA positive), human immunodeficiency virus (HIV) infection;
* Any clinically serious gastrointestinal dysfunction that may affect the intake, transport or absorption of the study drug, such as inability to take it orally Drugs, uncontrollable nausea and vomiting, history of extensive gastrointestinal resection, uncured recurrent diarrhea, atrophic gastritis (with The age of the disease is less than 60 years old), and the proton pump inhibitors (omeprazole, lansoprazole, pantoprazole, Rabeprazole, etc.) of stomach diseases, Crohn's disease, ulcerative colitis;
* Meet any of the following cardiac examination or disease standards:

  1. In the resting state, the average corrected QT interval (QTc) obtained from ECG examination, QTc interval>470 msec (QTcF=QT/RR1/3, when an abnormality is found in the first inspection, repeat the test twice within 48 hours, with an average of 3 times result calculation);
  2. Various abnormalities of heart rhythm, conduction, and resting ECG with serious clinical significance, such as complete left bundle branch block,

     Ⅲ degree conduction block, Ⅱ degree conduction block, PR interval>250 msec;
  3. Various factors that may increase the risk of QTc prolongation or the risk of arrhythmia events, such as heart failure, hypokalemia, Congenital long QT syndrome, first-degree relatives in family history have long QT syndrome or sudden death of unknown cause under 40 years old, Are using any drugs known to extend the QT interval;
* Left ventricular ejection fraction (LVEF) <50%;
* Have the following past history: interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid therapy;
* Acute onset or progressive, and the investigator believes that there are lung symptoms that are not suitable for enrollment or judged that interstitial Patients with high risk factors who are not suitable for entry into the group due to lung disease;
* Any serious or uncontrolled eye pathology, as judged by the investigator, may increase the safety risk of the patient, such as corneal ulcers, Bulbar conjunctivitis, etc.;
* The investigator determines that the patients are not suitable for participating in the study for other reasons (such as: the patient is unwilling to comply with the various procedures and limitations of the study). Regulations and requirements; those who have undergone allogeneic bone marrow transplantation; those who have other malignant tumors in the past 5 years or at the same time [excluding cervical cancer Cancer and treated basal cell carcinoma]; the patient's response to the active ingredients or inactive excipients of the test drug, chemical structure and research drug, medical history of hypersensitivity to similar drugs or similar drugs, etc.);
* At any time after the initial diagnosis, there is a confirmed EGFR 20 exon insertion mutation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
adverse event | through study completion, an average of 1.5 year
  Refers to adverse clinical events that occur during drug treatment, which may not have a causal relationship with the drug
Objective response rate (ORR) | through study completion, an average of 1.5 year
  According to the RECIST 1.1 standard, the best overall response (BOR) observed after enrollment of subjects is the proportion of subjects with complete remission (CR) or partial remission (PR)
Progression-free survival (PFS) | through study completion, an average of 1.5 year
  The time from the time a subject receives the first study treatment to the appearance of disease progression or death from any cause (whichever occurs first).
blood routine | through study completion, an average of 1.5 year
  the amount of red blood cell.
blood routine | through study completion, an average of 1.5 year
  the amount of white cell.
blood routine | through study completion, an average of 1.5 year
  the amount of platelet.

CONTACTS AND LOCATIONS:
Overall Officials: yuankai Shi, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (5):
- China (5):
  - Cancer hospital Chinese academy of medical sciences, Beijing, Beijing Municipality
  - Beijing cancer hospital, Beijing, Beijing Municipality
  - Henan university of science and technology first hospital, Luoyang, Henan
  - Henan cancer hospital, Zhengzhou, Henan
  - Hunan cancer hospital, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No